CLINICAL TRIAL: NCT06691074
Title: Systematic Assessment of the Acute Cavo-Tricuspid Isthmus Block Durability After Pulsed Electric Field Ablation
Brief Title: Cavo-Tricuspid Isthmus Block Durability After Pulsed Electric Field Ablation
Acronym: SECTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Predrag Stojadinovic, Medical Doctor, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28518/24; A-24-24; SECTION trial (Registry Identifier: SECTION)
Record Dates: First submitted 2024-09-16; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Flutter, Atrial; Cavotricuspid Isthmus Dependent Right Atrial Flutter; Catheter Ablation
Keywords: Pulsed Electric Field; Cavo-tricuspid Isthmus; Biderectional Block
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flower configuration (Active Comparator): Ablation of the CTI using a Farapulse catheter in flower configuration
  Interventions: Procedure: Catheter ablation of cavotricuspid isthmus using flower configuration of the Farapulse catheter
- Basket configuration (Active Comparator): Ablation of the CTI using a Farapulse catheter in basket configuration
  Interventions: Procedure: Catheter ablation of cavotricuspid isthmus using basket configuration of the Farapulse catheter

INTERVENTIONS:
Procedure: Catheter ablation of cavotricuspid isthmus using flower configuration of the Farapulse catheter — catheter ablation
  Arms: Flower configuration
Procedure: Catheter ablation of cavotricuspid isthmus using basket configuration of the Farapulse catheter — Catheter ablation of cavotricuspid isthmus using basket configuration of the Farapulse catheter
  Arms: Basket configuration

SUMMARY:
This study seeks to assess the acute durability of the CTI block when PEF energy is used. Second goal is to establish the optimal waiting time for the conduction recovery after PEF CTI ablation and to assess the utility of routine adenosine testing for dormant conduction. Moreover, this study aims to investigate the differences in acute efficacy and adverse events (hemolysis, coronary vasospasm) between the two available configurations (basket or flower) of the pentaspline Farawave catheter (Farapulse-Boston Scientific Inc, USA).

DETAILED DESCRIPTION:
Background Cavo-tricuspid isthmus (CTI) ablation is commonly performed as a concomitant procedure in patients undergoing pulmonary vein isolation (PVI) or more extensive left atrial ablations for the treatment of atrial fibrillation (AF). While the acute and long-term resumption of conduction in the CTI after radiofrequency ablation has already been investigated, the acute durability of the CTI block created by pulsed-electric field (PEF) energy has not been systematically evaluated.

Study population A prospective, multicentric randomized study conducted at high-volume centre with the routine use of intracardiac echocardiography (ICE). A total of 150 consecutive patients with paroxysmal AF undergoing PVI by PEF energy with documented typical atrial flutter or patients with persistent AF in whom catheter ablation of CTI is planned as a part of a complex procedure will be enrolled in the study.

Methods Procedures will be performed under general anaesthesia (GA) or deep analgo-sedation and on uninterrupted anticoagulation. One decapolar catheter will be introduced into the coronary sinus (CS). A duodecapolar catheter will be placed in the right atrium around the tricuspid annulus. A single transseptal puncture will be performed under ICE guidance. After obtaining the left atrial (LA) access, the Faradrive sheath will be redrawn into the right atrium. Patient presenting with AF or other atrial arrhythmias at the beginning of the procedure will be cardioverted. Prior to initiating pulsed field ablation (PFA) on the CTI, sublingual nitrates will be administered in the form of two sprays of nitroglycerin at a dose of 0.30 mg per spray. The CTI ablation will be performed during regular atrial pacing from the proximal CS at a cycle length of 600 ms. Sequential applications of PEF energy will be delivered in an overlapping fashion from the tricuspid annulus to the inferior cava vein under ICE guidance. Patients will be randomized in a 1:1 ratio based on the configuration of the catheter used to achieve CTI block (basket vs. flower). In both groups, three applications will be deployed at each spot. If acute block is not achievable using the randomized configuration, patients will be ablated using the other configuration and any additional lesions per operator discretion to achieve acute block. After demonstrating the bidirectional CTI block with standard pacing maneuvers (differential pacing from duodecapolar catheter and proximal CS), the surface electrocardiogram (ECG) will be analyzed across all 12 leads to evaluate for the presence of ST segment elevation. The left atrial procedure will be then performed during regular atrial pacing from the proximal CS. An eventual conduction recovery over the CTI and the corresponding time since the last ablation on the CTI will be recorded. Dormant conduction over the CTI will be assessed using an I.V. bolus of 12-18 mg of adenosine during continuous atrial pacing immediately after the confirmation of the CTI block and at the end of the procedure. The total waiting time and number of PEF applications on the CTI will be documented. At the end of the procedure, additional PEF applications per operator discretion on the CTI will be delivered if needed.

Sample size While no clear data on comparison of different Farapulse configurations on CTI are available, with 150 patients in the trial at a given expected acute success rate of 85 % in basket configuration given our clinical experience and a noninferiority design, a noninferiority margin of 15% at a power level of 82% can be tested.

Plasmatic biomarkers Venous blood samples for the assessment of plasma biomarkers (free hemoglobin [fHb], lactate dehydrogenase [LDH], total bilirubin, and haptoglobin) will be collected at two time points: before the procedure (T1) and after CTI isolation before LA ablation (T2).

Clinical implications

1. Achieving CTI block at the beginning of the catheter ablation of AF may provide sufficient waiting time to verify the durability of the block on TCI and thus enhance the long-term clinical effect of the procedure.
2. An absence of adenosine-induced CTI reconnection immediately after the CTI block could predict the durability of block at the end of the procedure and obviate the need for prolonged waiting period.
3. The use of the flower configuration to achieve CTI block could be associated with a non-inferior acute success rate and lower incidence of hemolysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with paroxysmal AF undergoing PVI by PEF energy with documented typical atrial flutter or patients with persistent AF in whom catheter ablation of CTI is planned as a part of a complex procedure
* Age ≥ 18 years at the time of study enrollment
* Signed informed consent

Exclusion Criteria:

* - LA diameter > 65 mm (measured in the parasternal long-axis view)
* History of CTI ablation in the past
* History of cardiac valve surgery
* Significant valvular defect
* Age below 18 years
* Pregnancy, breastfeeding
* Any disease with a life expectancy <1 year
* Uncorrected congenital heart disease or valvular obstruction
* Active myocarditis
* Untreated hypothyroidism or hyperthyroidism
* Recipient of any major organ transplant (e.g., lung, liver, heart)
* HIV positivity with a survival expectancy of less than five years due to HIV
* Chronic dialysis treatment
* Unwillingness to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The acute durability of the CTI block | During the ablation procedure
  The primary goal of this study is to assess the acute durability of the CTI block when PEF energy is used. The bidirectional block on the CTI will be demonstrated with standard pacing manoeuvres (differential pacing from duodecapolar catheter and proximal CS).

SECONDARY OUTCOMES:
The optimal waiting time for the conduction recovery after PEF CTI ablation | During the procedure
  Second goal is to establish the optimal waiting time for the conduction recovery after PEF CTI ablation.
The utility of routine adenosine testing for dormant conduction on the CTI | During the ablation procedure.
  Dormant conduction over the CTI will be assessed using an I.V. bolus of 12-18 mg of adenosine during continuous atrial pacing immediately after the confirmation of the CTI block and at the end of the procedure.
Concentration of plasma free haemoglobin | During the ablation procedure
  Plasma biomarker of hemolysis (free haemoglobin [fHb]) will be measured at two time points: before the procedure (T1) and after CTI isolation before LA ablation (T2). Levels of fHb will be compared among the study groups.
The presence of the coronary vasospasm | During the ablation procedure
  The surface electrocardiogram (ECG) will be analyzed across all 12 leads to evaluate for the presence of ST segment elevation (i.e. signs of the coronary vasospasm) after the CTI ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Morales G, Darrat YH, Lellouche N, Kim SM, Butt M, Bidwell K, Lippert W, Ogunbayo G, Hamon D, Di Biase L, Natale A, Parrott K, Elayi CS. Use of adenosine to shorten the post ablation waiting period for cavotricuspid isthmus-dependent atrial flutter. J Cardiovasc Electrophysiol. 2017 Aug;28(8):876-881. doi: 10.1111/jce.13233. Epub 2017 May 29. PMID 28429528
- [Background] Yoneda ZT, Shoemaker MB, Richardson T, Crawford D, Kanagasundram A, Shen S, Estrada JC, Holmes B, Lugo R, McHugh J, Saavedra P, Crossley G 3rd, Ellis CR, Montgomery JA, Michaud GF. Conduction Recovery After Cavotricuspid Isthmus Ablation When Performed With or Without Concomitant Atrial Fibrillation Ablation. JACC Clin Electrophysiol. 2020 Aug;6(8):989-996. doi: 10.1016/j.jacep.2020.04.031. PMID 32819535
- [Background] Chen J, de Chillou C, Ohm OJ, Hoff PI, Rossvoll O, Andronache M, Sadoul N, Magnin-Poull I, Erga KS, Aliot E. Acute resumption of conduction in the cavotricuspid isthmus after catheter ablation in patients with common atrial flutter. Real-time evaluation and long-term follow-up. Europace. 2002 Jul;4(3):255-63. doi: 10.1053/eupc.2002.0243. PMID 12134971